CLINICAL TRIAL: NCT06707064
Title: A Parallel-Group Controlled Clinical Study to Evaluate the Efficacy of Self-Family-Environment Empowerment (SFEE) Diet Management Intervention in Improving Outcomes for Pregnant Women With Gestational Diabetes Mellitus
Brief Title: SFEE Diet Management for Gestational Diabetes Mellitus
Acronym: SFEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ji Jing (Other)
Responsible Party: Sponsor-Investigator, Ji Jing, Head of Nurse Department, The First Affiliated Hospital of Shanxi Medical University
Organization: The First Affiliated Hospital of Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstShanxiMU2023; 2022-K205 (Other: Ethics Committee of the First Affiliated Hospital of Shanxi Medical University)
Record Dates: First submitted 2024-11-23; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational Diabetes Mellitus, SFEE Diet Management, Glycemic Control, Maternal Outcomes, Dietary Adherence
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the SFEE intervention group or a control group receiving standard dietary advice in a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to minimize bias during data collection and analysis. Participants and care providers were not masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFEE Diet Management Group ( Experimental Arm) (Experimental): Participants in this group received the Self-Family-Environment Empowerment (SFEE) diet management intervention, which included:
  Self-empowerment: Goal-setting, dietary planning, and evaluation. Family empowerment: Emotional support and supervision of dietary practices. Environmental empowerment: Peer group interaction, education, and support through WeChat groups.
  Routine nursing care was also provided alongside the intervention.
  Interventions: Behavioral: SFEE Diet Management Intervention
- Control Group (Active Comparator): Participants in this group received routine nursing care for gestational diabetes management, including:
  Medication guidance, dietary education using guidance charts, exercise plans, and self-monitoring.
  Dietary plans were customized based on individual patient needs, but no additional empowerment strategies (e.g., SFEE) were implemented.
  Interventions: Behavioral: Standard Dietary Advice

INTERVENTIONS:
Behavioral: SFEE Diet Management Intervention — A structured diet management program designed to improve glycemic control, dietary adherence, and maternal outcomes. It includes:
  Self-empowerment: Goal-setting, dietary planning, and evaluation. Family empowerment: Emotional support and supervision. Environmental empowerment: Peer group interaction and education via WeChat groups and in-person meetings.
  Arms: SFEE Diet Management Group ( Experimental Arm)
Behavioral: Standard Dietary Advice — Routine nursing care, including dietary education, exercise planning, and self-monitoring for gestational diabetes management.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the impact of the Self-Family-Environment Empowerment (SFEE) diet management intervention on glycemic control, maternal outcomes, and dietary adherence in pregnant women with gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a common complication of pregnancy, posing risks to maternal and fetal health. Effective management of GDM is critical to improving outcomes. This study aims to evaluate the potential of the Self-Family-Environment Empowerment (SFEE) diet management intervention in empowering pregnant women with GDM to improve glycemic control, dietary adherence, and maternal outcomes.

The study is conducted as a parallel-group controlled trial at the First Affiliated Hospital of Shanxi Medical University. Participants are allocated to two groups: an intervention group receiving routine care combined with the SFEE program and a control group receiving routine care only. The SFEE intervention integrates self-management strategies, family empowerment, and community learning, designed to support adherence to dietary recommendations and enhance participants' understanding of GDM management.

Primary outcomes include fasting blood glucose, postprandial glucose, and HbA1c levels measured after a 3-month intervention. Secondary outcomes include dietary adherence (assessed via a validated scale), GDM knowledge (measured using a questionnaire), and perceived social support (measured using the Perceived Social Support Scale)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gestational diabetes mellitus (GDM) based on the International Association of Diabetes and Pregnancy Study Groups (IADPSG) criteria.
* Aged 18-45 years.
* Pregnant women between 24-28 weeks of gestation at the time of enrollment.
* Able to provide informed consent.
* Access to a mobile phone and internet for study communication and follow-up.

Exclusion Criteria:

* Pregnant women with complications such as placental abruption, miscarriage, or induced abortion during the study period.
* Those unable to give informed consent or adhere to the intervention due to medical or personal reasons.
* History of severe medical conditions or other factors that might interfere with study participation (e.g., severe mental health conditions).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Glycemic Control (Fasting Blood Glucose Levels) | Baseline and 3 months post-intervention
  Change in fasting blood glucose levels (measured in mmol/L) from baseline to the end of the 3-month intervention period. This measure evaluates the effectiveness of the SFEE diet management intervention in improving blood glucose regulation in gestational diabetes mellitus.
Glycemic Control (HbA1c Levels) | Baseline and 3 months post-intervention
  Change in HbA1c levels (measured in %) from baseline to the end of the 3-month intervention period. This measure assesses the long-term blood sugar control improvements resulting from the SFEE diet management intervention compared to standard dietary advice.

SECONDARY OUTCOMES:
Dietary Adherence | Baseline and 3 months post-intervention
  Change in dietary adherence scores, measured using a validated adherence scale (range: 13-65, with higher scores indicating better adherence). This measure evaluates the participants' compliance with recommended dietary practices after the intervention.
GDM Knowledge | Baseline and 3 months post-intervention
  Change in gestational diabetes knowledge scores, measured using a validated questionnaire (range: 0-80, with higher scores indicating greater knowledge). This measure assesses the participants' understanding of gestational diabetes management, including diet and exercise.
Perceived Social Support | Baseline and 3 months post-intervention
  Change in perceived social support scores, measured using the Perceived Social Support Scale (range: 12-84, with higher scores indicating more support). This measure evaluates the impact of the intervention on participants' perceived emotional and social support.

CONTACTS AND LOCATIONS:
Overall Officials: Li Jun, Doctorate, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University
Locations (1):
- The First Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared as there is no provision for data sharing in the current study design, and ethical approval for data sharing has not been obtained. Researchers requiring data can contact the corresponding author for potential collaboration or data access requests in compliance with institutional and ethical guidelines

REFERENCES:
- See also: First Hospital of Shanxi Medical University Research — https://www.sydyy.com/
- Available data/document: Study Protocol: 2022-K205 — https://www.sydyy.com/ — The study protocol includes detailed methods, intervention description, and outcome measures. It is available upon reasonable request from the corresponding author.